CLINICAL TRIAL: NCT02042521
Title: A Dietary Supplement for Early Cigarette Withdrawal
Acronym: CIGAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Program Head, Neurochemical Imaging for Mood Disorders, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 021 / 2013
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Nicotine Dependence, Cigarettes, With Withdrawal
Keywords: Cigarette; Withdrawal; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Smokers (Active then Placebo) (Experimental): Healthy individuals who smokes at least 20 cigarettes per day
  Interventions: Dietary Supplement, Lactose Placebo
  Interventions: Drug: Dietary Supplement; Drug: Lactose Placebo
- Healthy Smokers (Placebo then Active) (Experimental): Healthy individuals who smokes at least 20 cigarettes per day
  Interventions: Dietary Supplement, Lactose Placebo
  Interventions: Drug: Dietary Supplement; Drug: Lactose Placebo

INTERVENTIONS:
Drug: Dietary Supplement — The active evening dietary supplement is taken at 22:00. The active morning dietary supplement is taken at 8:00-8:15. The active evening dietary supplement is taken first. The active morning and evening dietary supplements are taken within 12 hours in time points as specified above.
Drug: Lactose Placebo — This research study involves a placebo dietary supplement that does not have any of or only partial of the active ingredients in the active dietary supplement. The placebo dietary supplement will be given in identical time points to match that of the active dietary supplements.
  Other Names: Placebo

SUMMARY:
The purpose of this study is to determine whether a dietary supplement (DS) is effective in protecting against sad mood during early cigarette withdrawal. This study will also assess whether the dietary supplement will be well tolerated during early cigarette withdrawal.

DETAILED DESCRIPTION:
100 subjects who smoke at least 20 cigarettes per day will come in on two different days, at least one week apart, in a randomized, double blind, within subject, placebo controlled design. On each day subjects will refrain from smoking cigarettes for 8 hours. On one day subjects will take the active DS (taken in two doses, the evening dose is taken at 22:00 of the night before the test day and the morning dose is taken at 8:00 of the test day) and on the other day subjects will take placebo (also taken in two doses at the same time points of the active DS). Mood symptoms and symptoms of cigarette withdrawal will be compared across the two different days. Measures of mood symptom monitoring will include self report on a scale of 1 to 10, standardized rater questions about mood, and 6 hours into withdrawal, a standardized mood induction will be done with mood assessment. Symptoms of cigarette withdrawal will be assessed over the duration of withdrawal with applied standardized rating scales by trained raters. For the first 15 - 30 subjects, on each day, a health assessment of a physical exam and blood work will be completed at the end of the withdrawal period on both test days as well as for the initial assessment appointment.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* age 18-65
* generally good physical health
* not using any illicit substances
* smoke on average at least 20 cigarettes/day.

Exclusion Criteria:

* Recent history of myocardial infarction and / or stroke
* active substance abuse except for nicotine and active fluctuant medical conditions. (present and ongoing within 3 months)
* Score of higher than 7 on the 17- item Hamilton Depression Rating Scale
* Positive results for the pregnancy testing done on the first assessment visit.
* A specific allergy to fruit-based ingredient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in the Visual Analog Scale as Compared to Baseline Compared Across Two Conditions | Two sessions at least one week apart
  VAS uses a 10-cm scale for participants to indicate the extent to which each of them feel happy or sad. The change in VAS before versus after sad mood induction is the change score in VAS. The change score on the day with active dietary supplement is compared to the change score on the day with the placebo dietary supplement.

SECONDARY OUTCOMES:
Potential Side Effects Questionnaire | Twice on both test days: once in the morning right before the morning active or placebo dietary supplement and once more right after the observed break
  Structured questionnaires to assess the potential occurrence of side effects from Component A and Component B of the DS. In general, reported Component A side effects are fairly minor. Some of the reported side effects include nausea, headaches, fatigue, heartburn and joint pain. Reported side effects with Component B include: drowsiness, nausea and headaches, dizziness, fatigue, and lethargy
Profile of Mood States | Anytime during initial assessment visit. On both test days, at least 1 week apart at: (7:35-8:00); (8:40-9:05); (11:20-11:45); (12:25-12:50); (13:10-13:30); (14:30-14:55)
  The POMS contains 65 adjectives rated by participants on a 5-point scale. Six factors are derived that include tension, depression, anger, fatigue, vigor and confusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Meyer, MD, PhD, Principal Investigator — Research Imaging Centre, Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca/research